CLINICAL TRIAL: NCT03310073
Title: Immunogenicity and Safety Profile of Primary Dose of Bivalent OPV (bOPV Bio Farma) Given Simultaneously With Pentabio® And Inactivated Poliovirus Vaccine (IPV) at the 4th Visit in Indonesian Infants
Brief Title: Immunogenicity and Safety Profile of Primary Dose of bOPV Bio Farma Given Simultaneously With Pentabio And IPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bOPV 0416
Record Dates: First submitted 2017-04-05; First posted 2017-10-16 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bOPV (bivalent OPV Bio Farma) (Experimental): bOPV one dose corresponds to 2 drops (0.1ml). The vaccine shall be given orally.
  The subject received bOPV, Pentabio and IPV according to the study schedule.
  Interventions: Biological: bOPV; Biological: Pentabio; Biological: IPV

INTERVENTIONS:
Biological: bOPV — Batch Number: 2042015
  Other Names: bivalent Oral Polio Vaccine
Biological: Pentabio — Batch number: 5050115 The vaccine shall be given intramuscularly.
  Other Names: DTP-HB-Hib Vaccine
Biological: IPV — The vaccine shall be given intramuscularly.

SUMMARY:
This study is to assess protectivity following four doses of bOPV which given simultaneously with Pentabio® and 1 dose of IPV at the 4th visit

DETAILED DESCRIPTION:
To describe serological response after four doses of bOPV with 1 dose of IPV. To describe the antibody status to polio 60 days after birth dose of bOPV To assess the safety of bOPV which given simultaneously with Pentabio® and 1 dose 1 dosde of IPV at the 4th visit

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full term, newborns infants.
* Newborns residing within a relatively short and easily accessible distance (<30 km) from the study clinic(s) and not planning to travel away during the entire study period.
* Infant born after 37 weeks of pregnancy
* Infant weighing 2.5 kg or more at birth (Birth weight > 2.5 kg)
* Healthy newborns, with no history of asphyxia or meconium aspiration.
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
* Parents will commit themselves to comply with the indications of the investigator and with the schedule of the trial.
* Mother at least elementary school graduate

Exclusion Criteria:

* Child concomitantly enrolled or scheduled to be enrolled in another trial
* Known history of congenital or acquired immunodeficiency (including HIV infection)
* Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature ≥ 37.5°C )
* Newborns requiring hospitalization at birth.
* Infant immunized with non-scheduled bOPV or IPV during trial

Ages: 1 Minute to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with anti polio titer ≥ 8 for type 1, 2 and type 3 | 30 days after the last vaccination
  Evaluate protectivity

SECONDARY OUTCOMES:
Percentage of infants with increasing antibody titer >= 4 times | 30 days after the last vaccination
  Serological response after four doses of bOPV with 1 dose of IPV
Percentage of infants with transition of seronegative to seropositive | 30 days after the last vaccination
  Serological response after four doses of bOPV with 1 dose of IPV
Geometric Mean Titer (GMT) after four doses of bOPV with 1 dose of IPV | 30 days after the last vaccination
  Geometric Mean Titer (GMT) 30 days after the last vaccination
Number and severity of systemic adverse events (AEs) after each dose of bOPV, which given simultaneously with Pentabio and 1 dose of IPV | first 30 minutes, 24hour, 48hour, 72hour and 30 days after vaccination.
  Assess the safety of bOPV
Number of serious adverse events (SAE) which occured during the study | 30 days after the last vaccination
  Assess the safety of bOPV

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, Principal Investigator — Hasan Sadikin General Hospital
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia